CLINICAL TRIAL: NCT06544278
Title: Evaluation of the Effects of Probiotics on Sperm Quality in Middle-aged Men: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: The Impact of Probiotics on Sperm Quality in Middle-aged Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2023010
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Sperm Quality
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double(Participant,Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Participants in the probiotic group received 1 sachet probiotic product per day.
  Interventions: Dietary Supplement: probiotic product
- Placebo group (Placebo Comparator): Participants in the placebo group received 3g of maltodextrin per day.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: probiotic product — During the experiment, subjects take one sachet probiotic product daily. Evaluation is conducted by monitoring the subjects' semen concentration before and after this trial.
  Arms: Probiotic group
Dietary Supplement: Maltodextrin — During the experiment, subjects take one sachet maltodextrin daily with 3.0g. Evaluation is conducted by monitoring the subjects' semen concentration before and after this trial.
  Arms: Placebo group

SUMMARY:
The clinical trial aims to investigate the impact of probiotic strain BL21 on sperm quality among 46 middle-aged male participants. The primary objective is to validate whether probiotic strain BL21 can effectively improve sperm quality among middle-aged male participants. Initially, participants were instructed to consume the recommended amount of probiotic powder for approximately 8 weeks. At baseline, week 4, and week 8 endpoints, semen analysis, hormone level testing, serum cytokine testing were conducted on the participants, and stool samples were collected from them.

DETAILED DESCRIPTION:
Research has indicated that an increase in male age is independently associated with a reduction in the percentage of motile sperm and sperm with normal morphology, especially in men over 40 years old, potentially linking to a decline in fertility rates. Preclinical studies have shown that supplementation with Long Bifidobacterium can regulate immune responses, inhibit tissue inflammatory factors, and the predictive functions of the gut microbiota suggest an increase in gene abundance within pathways related to secondary metabolite production, antibiotic synthesis, and amino acid biosynthesis in the gut microbiota. To ascertain the effectiveness of the Bifidobacterium BL21 product, a consumer testing experiment was conducted by the investigators to evaluate and gather data on alterations in the gut microbiota of participants prior to and following the use of the product. The trial spanned over 8 weeks, with washout periods incorporated at the commencement and conclusion. Throughout the study, participants ingested Bifidobacterium BL21 and were subjected to a series of health examinations and assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 40-59 years old.
2. Normal levels of gonadotropins, testosterone, and serum prolactin.
3. No use of other traditional Chinese and Western medicines for oligoasthenoteratozoospermia treatment in the past 3 months.
4. Patients who can understand the clinical study and commit to complying with the study requirements and procedures.
5. Patients who have signed the informed consent form and are able to complete the study as per the trial protocol.

Exclusion Criteria:

1. Organic lesions of the reproductive system;
2. Use of antibiotics in the two weeks prior to recruitment;
3. Sexual dysfunctions such as erectile dysfunction, ejaculatory abnormalities, preventing completion of sexual intercourse;
4. Genitourinary infections, such as Chlamydia or Mycoplasma infections;
5. Abnormal sex hormone levels;
6. Obesity (BMI greater than 28);
7. History of allergies to the probiotic preparations used in this study;
8. Severe cardiovascular or cerebrovascular diseases, liver or kidney dysfunction, hematologic disorders, psychiatric illnesses, or other severe comorbidities;
9. Use of medications in the past 3 months that may affect the trial;
10. According to the investigator's judgment, the subject's condition does not qualify them for participation in the study.

Ages: 40 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sperm Motility Percentage Assessed by Computer-Assisted Sperm Analysis System (CASA) After 8 Weeks | 8 weeks
  The percentage change in sperm motility will be measured using a Computer-Assisted Sperm Analysis System (CASA). Sperm samples will be collected at baseline and after the 8-week intervention. Results will be presented as mean ± standard deviation. The data will be used to assess the effect of Bifidobacterium longum subsp. longum BL21 on sperm motility in middle-aged men.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shangdong University, Jinan, Shangdong, China

IPD SHARING:
Plan to Share IPD: No